CLINICAL TRIAL: NCT03489343
Title: A Phase 1, Open-Label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Antineoplastic Activity of Sym023 (Anti-TIM-3) in Patients With Advanced Solid Tumor Malignancies or Lymphomas
Brief Title: Sym023 (Anti-TIM-3) in Patients With Advanced Solid Tumor Malignancies or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym023-01
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Cancer; Solid Tumor; Lymphoma
Keywords: Locally advanced/unresectable; Metastatic solid tumor; Lymphoma; Anti-TIM-3; TIM-3; TIM3
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Sym023 0.03 mg/kg (Experimental): Sym023 was administered at a dose of 0.03 mg/kg by intravenous infusion
  Interventions: Drug: Sym023
- Sym023 0.1 mg/kg (Experimental): Sym023 was administered at a dose of 0.1 mg/kg by intravenous infusion
  Interventions: Drug: Sym023
- Sym023 0.3 mg/kg (Experimental): Sym023 was administered at a dose of 0.3 mg/kg by intravenous infusion
  Interventions: Drug: Sym023
- Sym023 1.0 mg/kg (Experimental): Sym023 was administered at a dose of 1.0 mg/kg by intravenous infusion
  Interventions: Drug: Sym023
- Sym023 3.0 mg/kg (Experimental): Sym023 was administered at a dose of 3.0 mg/kg by intravenous infusion
  Interventions: Drug: Sym023
- Sym023 10.0 mg/kg (Experimental): Sym023 was administered at a dose of 10.0 mg/kg by intravenous infusion
  Interventions: Drug: Sym023
- Sym023 20.0 mg/kg (Experimental): Sym023 was administered at a dose of 20.0 mg/kg by intravenous infusion
  Interventions: Drug: Sym023

INTERVENTIONS:
Drug: Sym023 — Sym023 is a recombinant, fully human antibody that binds TIM-3 and induces activation of immune cells.
  Other Names: Anti-TIM-3

SUMMARY:
This was the first study to test Sym023 in humans. The primary purpose of this study was to see if Sym023 is safe and tolerable for patients with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available.

DETAILED DESCRIPTION:
This study evaluated the preliminary safety, tolerability, and dose-limiting toxicities (DLTs) of Sym023, a recombinant, fully human, anti-T-cell immunoglobulin and mucin-domain containing-3 (anti-TIM-3) monoclonal antibody (mAb). The goal was to establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of sequential escalating doses of Sym023 when administered once every 2 weeks (Q2W) by intravenous (IV) infusion to patient cohorts with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available. If an MTD was not identified, a maximum administered dose (MAD) was to be determined. Sym023 was given to patients in escalating dose cohorts; each patient was given one fixed dose level.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age at the time of obtaining informed consent.
* Documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic; patients with documented lymphomas.
* Malignancy (solid tumor or lymphoma) that is currently not amenable to surgical intervention due to either medical contraindications or nonresectability of the tumor.
* Refractory to or intolerant of existing therapy(ies) known to provide clinical benefit.
* Measurable or non-measurable disease according to RECIST v1.1 or RECIL 2017.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Not of childbearing potential or who agree to use a highly effective method of contraception during the study beginning within 2 weeks prior to the first dose and continuing until 6 months after the last dose of study drug.

Exclusion Criteria:

* Women who are pregnant or lactating, or intending to become pregnant before, during, or within 6 months after the last dose of study drug. Women of childbearing potential (WOCBP) and fertile men with WOCBP-partner(s) not using and not willing to use a highly effective method of contraception.
* Known, untreated central nervous system (CNS) or leptomeningeal metastases, or spinal cord compression, patients with any of the above not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
* Hematologic malignancies other than lymphomas.
* Active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to Cycle 1/Day 1 (C1/D1) unless adequately treated and considered stable.
* Active uncontrolled bleeding or a known bleeding diathesis.
* Clinically significant cardiovascular disease or condition.
* Significant ocular disease or condition, including history of autoimmune or inflammatory disorder.
* Significant pulmonary disease or condition.
* Current or recent (within 6 months) significant gastrointestinal (GI) disease or condition.
* An active, known, or suspected autoimmune disease, or a documented history of autoimmune disease or syndrome, requiring systemic steroids or other immunosuppressive medications.
* History of significant toxicities associated with previous administration of immune checkpoint inhibitors that necessitated permanent discontinuation of that therapy.
* Patients with unresolved > Grade 1 toxicity associated with any prior antineoplastic therapy, with exceptions.
* Inadequate recovery from any prior surgical procedure, or having undergone any major surgical procedure within 4 weeks prior to C1/D1.
* Known history of human immunodeficiency virus (HIV) or known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, FRCPC, Principal Investigator — Princess Margaret Cancer Centre
Locations (4):
- United States (3):
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sym023 0.03 mg/kg: Sym023 0.03 mg/kg intravenous infusion once every 2 weeks
- Sym023 0.1 mg/kg: Sym023 0.1 mg/kg intravenous infusion once every 2 weeks
- Sym023 0.3 mg/kg: Sym023 0.3 mg/kg intravenous infusion once every 2 weeks
- Sym023 1.0 mg/kg: Sym023 1.0 mg/kg intravenous infusion once every 2 weeks
- Sym023 3.0 mg/kg: Sym023 3.0 mg/kg intravenous infusion once every 2 weeks
- Sym023 10.0 mg/kg: Sym023 10.0 mg/kg intravenous infusion once every 2 weeks
- Sym023 20.0 mg/kg: Sym023 20.0 mg/kg intravenous infusion once every 2 weeks
Period: Overall Study
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Started | 1 | 1 | 3 | 3 | 3 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 3 | 7 | 6
Not completed — Documented progressive disease | 1 | 0 | 3 | 1 | 3 | 5 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Clinical progression | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised all consented patients who had received at least a fraction of 1 dose of study drug. The patients in the FAS contributed to the analyses as allocated to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 1 | 1 | 5 | 5 | 16
  >=65 years | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 8
Age, Continuous [Median (Full Range); unit: years] | 64 [64 to 64] | 64 [64 to 64] | 62 [59 to 67] | 66 [45 to 70] | 71 [59 to 72] | 54 [37 to 76] | 61 [36 to 74] | 63 [36 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 3 | 4 | 4 | 16
  Male | 1 | 0 | 1 | 1 | 0 | 3 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 3 | 3 | 2 | 7 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
  White | 1 | 1 | 3 | 3 | 2 | 2 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5
  United States | 1 | 1 | 3 | 2 | 2 | 5 | 5 | 19
ECOG PS [Count of Participants; unit: Participants] — The ECOG PS is Eastern Cooperative Oncology Group performance status, and is a measure of how well a person is able to carry out ordinary daily activities while living with cancer, and provides an estimate of what treatments a person may tolerate. It has scores ranging from 0 to 5 with 0 being best and 5 being worst. ECOG is commonly used as a prognostic tool, as a selection criterion for cancer research, and to help determine treatment. Patients with an ECOG PS of 0 or 1 were included in the trial.
  Participants
    1 | 1 | 1 | 2 | 2 | 3 | 6 | 4 | 19
    0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Treatment Emergent Adverse Events (AEs) Meeting Dose-limiting Toxicity (DLT) Criteria.
Description: Assess the safety and tolerability of Sym023 on a Q2W (once every 2 weeks) schedule to establish the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D). Assessment based on the occurrence of AEs meeting DLT criteria measured during Cycle 1. The MTD was to be determined by those DLTs that occurred during C1 in either more than 1 patient in a 3 to 6 patient cohort or ≥33.3% of patients in the event of an expanded 7 to 12 patient cohort. One patient in the 10.0 mg/kg dose cohort was not evaluable for MTD as she did not complete C1 for a reason other than drug toxicity (i.e., discontinuation after 1 dose due to patient withdrawal of consent). However, this patient was included in the evaluation of other outcomes.
Time Frame: 28 days
Population: DLT analysis set of patients who completed treatment dosing in a 4-week (28 day) period that was Cycle 1. One patient out of 7 patients in Group 10mg/kg did not complete Cycle 1 and are not included in the "participants analyzed"
Measure: Number; unit: Number of DLTs
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 6
Number of DLTs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Evaluation of the Immunogenicity of Sym023.
Description: Serum sampling to assess the potential for anti-drug antibody (ADA) formation. The number of patients with positive samples at indicated visits is presented.
Time Frame: Baseline up to 6-months follow-up, approximately 1 year
Population: Full analysis set of all randomised and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 6
Participants
  Cycle 1 days 1 and 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 days 1 and 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 days 1 and 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 5 day 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Cycle 6 day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 7 day 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  End of treatment | 0 | 1 | 1 | 1 | 0 | 0 | 0
  1-month follow up | 0 | 1 | 1 | 1 | 0 | 0 | 0
  3-month follow up | 0 | 0 | 0 | 1 | 0 | 0 | 0

3. Secondary Outcome: Evaluation of Objective Response (OR) or Stable Disease (SD) by RECIST v1.1
Description: OR or SD Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). The number of patients with confirmed or unconfirmed OR (partial or complete response) is presented. Duration of SD for patients with best overall response = SD was defined as the time from the day of first study treatment to the start of radiologic disease progression or death. If the patient did not have a radiological disease progression or death, the duration of SD was defined as the time from the day of first study treatment to the date of the last SD assessment.
Time Frame: 24 months
Population: Full analysis set of randomised and treated patients who was evaluable for response. One patient out of 7 in group 10mg/kg was not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 6
Participants
  OR rate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD >16 weeks | 0 | 1 | 0 | 0 | 0 | 0 | 2
  SD ≤16 weeks | 0 | 0 | 0 | 2 | 2 | 0 | 3

4. Secondary Outcome: Evaluation of Objective Response (OR) or Stable Disease (SD) by iRECIST
Description: OR or SD Assessed by Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST). The number of patients with confirmed or unconfirmed OR (partial or complete response) is presented. Duration of SD for patients with best overall response = SD was defined as the time from the day of first study treatment to the start of radiologic disease progression or death. If the patient did not have a radiological disease progression or death, the duration of SD was defined as the time from the day of first study treatment to the date of the last SD assessment.
Time Frame: 24 months
Population: Full analysis set of randomised and treated patients who were evaluable for response. One patient out of 7 in group 10mg/kg was not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 6
Participants
  OR rate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  iSD >16 weeks | 0 | 1 | 0 | 1 | 1 | 0 | 1
  iSD ≤16 weeks | 0 | 0 | 0 | 2 | 1 | 0 | 4

5. Secondary Outcome: Evaluation of Objective Response (OR) or Stable Disease (SD) by RECIL 2017.
Description: OR or SD Assessed by Response Evaluation Criteria in Lymphomas 2017 (RECIL 2017)
Time Frame: 24 months
Population: No lymphomas were recorded in this trial, therefore it was not possible to do the RECIL evaluation.
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Time to Progression (TTP) of Disease.
Description: Based on time of enrollment to first evidence of progression on imaging studies, as assessed by RECIST v1.1, RECIL 2017, or iRECIST, depending on tumor type. The numbers shown below correspond to the values related to RECIST v1.1.
Time Frame: 24 months
Population: The full analysis set of randomized and treated patients who were evaluable for response. One patient out of 7 in group 10mg/kg was not evaluable for response or time to progression (TTP) as the patient left trial due to Adverse Event
Measure: Median (Full Range); unit: months
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 6 | 6
months | 1.81 [1.81 to 1.81] | 7.89 [7.89 to 7.89] | 1.18 [0.72 to 1.38] | 3.48 [1.87 to 3.55] | 1.28 [1.12 to 3.52] | 1.68 [0.03 to 2.07] | 5.36 [1.61 to 5.55]

7. Secondary Outcome: Area Under the Concentration-time Curve in a Dosing Interval (AUC).
Description: The AUC after first dose was estimated using non-compartmental methods. Blood samples for PK analysis were taken at the following timepoints: before the start of the infusion, at the end of the infusion and at 2, 4, 8, 24, 48 and 168 hours after the end of the infusion. Actual timepoints were recorded.
Time Frame: From before the start of the infusion to 168 hours after the end of the infusion
Population: Pharmacokinetic analysis set (same as the full analysis set) of all randomised and treated patients
Measure: Mean (Full Range); unit: h*μg/mL
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 6
h*μg/mL | 70 [70 to 70] | 176 [176 to 176] | 878 [680 to 1158] | 3193 [2449 to 4194] | 8062 [4498 to 12358] | 30581 [7039 to 45928] | 77262 [54275 to 85463]

8. Secondary Outcome: Maximum Concentration (Cmax)
Description: Outcome measure after first dose was derived from observed data. Blood samples for PK analysis were taken at the following timepoints: before the start of the infusion, at the end of the infusion and at 2, 4, 8, 24, 48 and 168 hours after the end of the infusion. Actual timepoints were recorded.
Time Frame: From before the start of the infusion to 168 hours after the end of the infusion
Population: Pharmacokinetic analysis set (same as the full analysis set) of all randomised and treated patients
Measure: Mean (Full Range); unit: μg/mL
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 6
μg/mL | 0.85 [0.85 to 0.85] | 1.98 [1.98 to 1.98] | 7.94 [5.67 to 11.56] | 23.71 [19.87 to 28.30] | 68.03 [52.88 to 84.16] | 232.11 [183.26 to 288.01] | 470.24 [294.82 to 543.46]

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax)
Description: as for outcome 8
Time Frame: From before the start of the infusion to 168 hours after the end of the infusion
Population: Pharmacokinetic analysis set (same as the full analysis set) of all randomised and treated patients
Measure: Mean (Full Range); unit: hours
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 7 | 6
hours | 4.5 [4.5 to 4.5] | 0.6 [0.6 to 0.6] | 1.2 [0.5 to 2.5] | 4.5 [4.4 to 4.7] | 1.8 [0.6 to 2.6] | 3.4 [0.5 to 8.5] | 7.3 [0.5 to 20.8]

10. Secondary Outcome: Trough Concentration (Ctrough)
Description: as for outcome 8
Time Frame: From before the start of the infusion to 168 hours after the end of the infusion
Population: Pharmacokinetic analysis set (same as the full analysis set) of all randomized and treated patients. Data for cohort 0.03mg/kg: Ctrough at 168 hours were below the limit of quantification, hence no reported data
Measure: Mean (Full Range); unit: μg/mL
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 5 | 6
μg/mL | NA [NA to NA] — Ctrough at 168 hours were below the limit of quantification, hence no reported data | 0.16 [0.16 to 0.16] | 1.26 [0.76 to 1.85] | 6.39 [4.26 to 9.37] | 12.88 [4.09 to 26.10] | 74.33 [37.47 to 116.52] | 146.96 [101.68 to 189.29]

11. Secondary Outcome: Terminal Elimination Half-life (T½)
Description: Outcome measure after first dose was estimated using non-compartmental methods. Blood samples for PK analysis were taken at the following timepoints: before the start of the infusion, at the end of the infusion and at 2, 4, 8, 24, 48 and 168 hours after the end of the infusion. Actual timepoints were recorded.
Time Frame: From before the start of the infusion to 168 hours after the end of the infusion
Population: Pharmacokinetic analysis set (same as the full analysis set) of all randomised and treated patients. Data for cohort 0.03mg/kg: T½ could not be accurately calculated due to few datapoint within the elimination period
Measure: Mean (Full Range); unit: hours
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 0 | 2 | 2 | 1
hours | NA — T½ could not be accurately calculated due to few datapoints within the elimination | 105.10 [105.10 to 105.10] | 153.49 [136.70 to 164.11] |  | 140.60 [112.78 to 168.42] | 185.22 [153.43 to 217.01] | 203.07 [203.07 to 203.07]

12. Secondary Outcome: Clearance (CL)
Description: as for outcome 11
Time Frame: From before the start of the infusion to 168 hours after the end of the infusion
Population: Pharmacokinetic analysis set (same as the full analysis set) of all randomized and treated patients. Data for cohort 0.03mg/kg: Clearence could not be accurately calculated since too few datapoint within the elimination period
Measure: Mean (Full Range); unit: mL/h)/kg
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
Number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 0 | 0
mL/h)/kg |  | 0.501 [0.501 to 0.501] | 0.364 [0.364 to 0.364] |  | 0.582 [0.582 to 0.582] |  |

ADVERSE EVENTS:
Time Frame: 24 months
Description: Only treatment-emergent adverse events (AEs) are presented in clinicaltrials.gov, defined as AEs with onset dates on or after the first dose of study medication or AEs that occurred before the first dose of study medication and increased in severity after the first dose of study medication up to the last dose of study drug plus 30 days.
Arm/Group | Sym023 0.03 mg/kg | Sym023 0.1 mg/kg | Sym023 0.3 mg/kg | Sym023 1.0 mg/kg | Sym023 3.0 mg/kg | Sym023 10.0 mg/kg | Sym023 20.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 3/3 | 0/3 | 2/3 | 1/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/3 | 0/3 | 0/3 | 2/7 | 1/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 3/3 | 7/7 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sym023 0.03 mg/kg (N=1) | Sym023 0.1 mg/kg (N=1) | Sym023 0.3 mg/kg (N=3) | Sym023 1.0 mg/kg (N=3) | Sym023 3.0 mg/kg (N=3) | Sym023 10.0 mg/kg (N=7) | Sym023 20.0 mg/kg (N=6)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sym023 0.03 mg/kg (N=1) | Sym023 0.1 mg/kg (N=1) | Sym023 0.3 mg/kg (N=3) | Sym023 1.0 mg/kg (N=3) | Sym023 3.0 mg/kg (N=3) | Sym023 10.0 mg/kg (N=7) | Sym023 20.0 mg/kg (N=6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (4) | 2 (3) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Pyrexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03489343/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT03489343/SAP_001.pdf